CLINICAL TRIAL: NCT05019638
Title: Evaluating the Effectiveness of Local Multimodal Injection in Controlling Pain, Limiting Complications, and Reducing Cost as Compared to Regional Anesthesia for Treating Rotational Ankle Fractures.
Brief Title: Local Multimodal Injection Versus Regional Anesthesia in Controlling Pain for Treating Rotational Ankle Fractures
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 137271
Record Dates: First submitted 2021-07-19; First posted 2021-08-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ankle Fractures
Keywords: rotational ankle fractures; regional anesthesia; local multimodal injection; pain
MeSH Terms: conditions — Ankle Fractures; Pain | interventions — Bupivacaine; Epinephrine; Morphine; Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regional anesthesia group (Active Comparator): Standard single-shot anesthesia consists of bupivacaine 0.25% with epinephrine 1:400,000.
  Interventions: Drug: Regional anesthesia group
- Local multimodal analgesia group (Experimental): Local multimodal analgesia composition will include 5mg of morphine, 500 mg of epinephrine, 15mg of ketorolac, and 20mg of bupivacaine.
  Interventions: Drug: Local multimodal analgesia group

INTERVENTIONS:
Drug: Regional anesthesia group — bupivacaine 0.25% with epinephrine 1:400,000.
  Other Names: Marcaine (bupivacaine); Adrenalin (epinephrine)
  Arms: Regional anesthesia group
Drug: Local multimodal analgesia group — 5mg of morphine, 500 mg of epinephrine, 15mg of ketorolac, and 20mg of bupivacaine.
  Other Names: MS Contin, Astramorph, Depodur, Duramorph, Infumorph, Kadian, MorphaBond, Arymo ER (morphine); Adrenalin (epinephrine); Toradol (ketorolac); Marcaine (bupivacaine)
  Arms: Local multimodal analgesia group

SUMMARY:
The investigators plan to evaluate the efficacy in reducing post-operative pain between local multimodal analgesia as compared to regional anesthesia in rotational ankle fractures.

DETAILED DESCRIPTION:
Pain control is a chief domain in patient-centered care and may play a key role in outcome-driven reimbursement as a focus on payment strategies shifts in this direction. The Center for Medicaid and Medicare Services has developed the Total Performance Score for Hospitals, which is factored into the reimbursement for provided services. Pain Management is one of the main contributors to the score. Moreover, pain control has been shown to improve patient satisfaction, which is of increasing importance in medicine today.

The United States is in the midst of an opioid epidemic where we consume 80% of the world's narcotics with only 5% of the world's population. Prescription opioids may play a major role in up to 40% of opioid overdose deaths. Orthopedic surgeons are the top prescribing surgical specialists and the fourth-largest overall prescriber of narcotic medication, representing 7.7% of total opioid prescriptions. Given the magnitude and implications of the opioid epidemic, orthopedic surgeons have been tasked with delivering adequate pain control while avoiding excessive narcotic prescriptions that can lead to opioid addiction and opioid-related deaths.

Regional anesthesia has been extensively studied for operatively managed rotational ankle fractures. Foot and ankle surgery patients receiving regional anesthesia have been reported to have lower pain scores and less narcotic usage for up to 8 weeks post-operatively. In a prospective cohort study of ankle fracture patients, Investigators have demonstrated improved pain management in patients who received single-shot regional anesthesia as compared to control patients. In a blinded, prospective, randomized controlled trial, it was reported lower pain scores and longer analgesia in patients receiving peripheral nerve block as compared to control patients.

Local multimodal analgesia has been used extensively in the setting of total knee arthroplasty. Numerous studies have investigated the effect of these injections and shown a decrease in perioperative pain and the use of perioperative narcotics. A team of investigators looked at multimodal analgesia injections in femur fractures of all kinds. They found that in patients receiving the injection, their pain was decreased over the first postoperative day along with consuming fewer narcotics over the same time frame. Unfortunately, the randomization in this study resulted in an unequal distribution of injuries that may have biased the results. It was noted, "further investigations are required to establish the efficacy of this multimodal protocol for the individual surgical procedures considered."

Several aspects of the proposed study are innovative and the results of which will provide evidence for significant change. The proposed studies focuses on one of the most common skeletal injuries treated with surgical intervention by orthopaedic surgeons. These investigators are thus focusing on an area with widespread implications where a small change in practice could result in extensive change through the system. The overarching goal for this investigation is to optimize postoperative pain control delivery while limiting narcotic medication consumption.

There are currently no studies that compare the effectiveness and cost between local multimodal analgesia and regional anesthesia as it relates to rotational ankle fractures. Despite extensive use in arthroplasty, local multimodal analgesia has limited usage in the setting of fracture or acute injury. This represents a significant area of innovation and growth in the realm of orthopaedic traumatology. Given the commonplace nature of ankle fractures and the ability to perform regional anesthesia given the lack of compartment syndrome risk, these injuries represent the ideal candidate to explore a new mode of postoperative analgesia. Additionally, incorporating an anti-inflammatory medication into the local multimodal injection cocktail is novel. While a stigma associated with anti-inflammatory medications and impaired bone healing exist, single usage should be relatively low risk while providing significant local pain relief. The ability of local multimodal analgesia to provide similar pain control as regional anesthesia would expand the possibility of using local multimodal analgesia in locations that do not have an appropriately trained anesthesiologist for regional anesthesia. It may also improve the workflow and open the possibility of investigation as it relates to other common fractures.

The hypothesis is that ankle fracture patients with post-operative local multimodal analgesia will have similar Visual Analog Scale (VAS) pain scores as patients with post-operative regional anesthesia at 24 hours post-surgery. Secondary analyses will compare VAS pain scores at 1, 2, 4, and 8 hours post-operatively in addition to post-operative narcotic usage between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* isolated rotational ankle fracture
* operative intervention needed
* English or Spanish speaking
* provide informed consent
* able to communicate with the research team via email or phone

Exclusion Criteria:

* sustain concomitant head injury
* additional lower extremity fracture(s)
* open fracture
* prior drug dependency
* allergies to any of the ingredients in the local injection or peripheral nerve block
* any history of stroke
* major neurological deficit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | Pre-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 1-hour post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 2-hour post -operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 4-hour post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 8-hour post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 24-hour post-operative
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, MD, Principal Investigator — University of Utah Orthopaedics
Locations (2):
- United States (2):
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - University of Utah Orthopedics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No